CLINICAL TRIAL: NCT00339378
Title: Incidence and Mortality of Childhood Cancer Among Children of Farmer Pesticide Applicators
Brief Title: Incidence and Mortality of Childhood Cancer Among Children of Farmer Pesticide Applications
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999900025; OH00-E-N025
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-06-11

CONDITIONS: Pesticide Exposure
Keywords: Record Linkage; Retrospective; Cohort; Registries; Agricultural

SUMMARY:
Previous studies have estabished pesticide exposure as a possible risk factor for childhood cancer. The Agricultural Health Study (AHS), a prospective cohort study of pesticide exposure among 51,000 pesticide applicators in North Carolina and Iowa, provides an opportunity to study childhood cancer incidence and mortality among the children of pesticide applicators. Name and dates of birth for 21,985 children were previously provided by adult participants in the AHS. The current study seeks to identify cases of cancer among these children through record linkage to state cancer and death registries. Cancer incidence and mortality within the cohort will be compared with national data through standardized incidence and mortality ratios. A limited case-cohort comparison of pesticide exposures will also be performed. Approximately 44 cases of childhood cancer are expected to be identified. No follow-up or contact with cases is anticipated. It is anticipated that the study results will provide insight into the relationship of pesticide and other farm exposures to the pathogenesis of childhood cancer.

DETAILED DESCRIPTION:
Previous studies have estabished pesticide exposure as a possible risk factor for childhood cancer. The Agricultural Health Study (AHS), a prospective cohort study of pesticide exposure among 51,000 pesticide applicators in North Carolina and Iowa, provides an opportunity to study childhood cancer incidence and mortality among the children of pesticide applicators. Name and dates of birth for 21,985 children were previously provided by adult participants in the AHS. The current study seeks to identify cases of cancer among these children through record linkage to state cancer and death registries. Cancer incidence and mortality within the cohort will be compared with national data through standardized incidence and mortality ratios. A limited case-cohort comparison of pesticide exposures will also be performed. Approximately 44 cases of childhood cancer are expected to be identified. No follow-up or contact with cases is anticipated. It is anticipated that the study results will provide insight into the relationship of pesticide and other farm exposures to the pathogenesis of childhood cancer.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be included in the study if they are children of private pesticide applicators who participated in the AHS, and were born between 1975 and 1996.

EXCLUSION CRITERIA:

Subjects with age greater than 19 years during this period will be excluded as the outcome under study is childhood cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21985
Dates: Start 2000-06-28; Study Completion 2007-06-11

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - National Cancer Institute, Bethesda, Maryland
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina
  - Environmental Protection Agency, Research Triangle Park, North Carolina